CLINICAL TRIAL: NCT05945238
Title: Effect of Thrower's Ten Exercise Program on Shoulder Flexibility, Stability and Strength in Water Polo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Burak Asal, PT, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BU-ASAL-001
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Injuries
Keywords: Thrower's Ten; Water Polo; Flexibility; Stability; Strength
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrower's Ten (Experimental)
  Interventions: Other: Thrower's Ten Exercise Program
- Control (No Intervention)

INTERVENTIONS:
Other: Thrower's Ten Exercise Program — T10 group were given thrower's ten exercises 3 times per week for 10 weeks, each exercise being 2x10 repetitions.
  Arms: Thrower's Ten

SUMMARY:
Context: Studies have shown that the thrower's ten rehabilitation program is effective in the prevention and rehabilitation of injuries in overhead throwing sports. However its effect on water polo sports is still unknown.

Objective: To investigate the effect of thrower's ten (T10) exercise program on shoulder flexibility, stability and strength in water polo athletes.

Design: Randomized controlled clinical trial. Setting: Middle East Technical University swimming pool and training facilities.

Intervention(s): T10 group were given thrower's ten exercises 3 times per week for 10 weeks, each exercise being 2x10 repetitions. Athletes in the control group were not given any additional exercise to their weekly water polo training.

Main Outcome Measure(s): Before and after the exercise, the upper extremity internal and external rotation strength of the athletes was measured with isokinetic dynamometer, the shoulder stability was measured with the closed kinetic chain upper extremity test (CKCUEST), and the shoulder flexibility was measured with the help of the shoulder joint internal and external rotation motion flexibility test.

Key Words: Thrower's Ten, Water Polo, Stability, Flexibility, Strength

DETAILED DESCRIPTION:
Before starting the study, individuals were informed about the purpose of the study, the test protocols to be applied and the program.

Individuals who met the inclusion criteria were randomly allocated into two groups named T10 (n=24) and Control (n=26) in a single blinded manner using a computer-based online site called "Random Lists". Three separate evaluation tests were administered before and 10 weeks after the start of the study.

Individuals in the T10 group underwent T10 exercise program with a physiotherapist or trainer for 10 weeks with 3 sessions per week and at least 1 day between sessions. Individuals in the control group were followed up for 10 weeks as they continued their weekly team training without being actively subjected to an extra program., After the inital evaluations were completed in the T10 group, exercises were started 1 week before the study and the exercises were taught. Elastic resistance band in the appropriate color to be used in the program were determined based on 70% difficulty according to the OMNI scale.

The athletes participating in the study were evaluated twice in total, at the beginning and at the end of the study. Sociodemographic data including age, weight, height, gender, BMI and dominant side were collected. Shoulder strength of the participants was evaluated with an isokinetic dynamometer in 90° abduction with external and internal rotation force test at angular velocities of 60°/s and 180°/s in two different ways. Upper extremity stability of the participants was evaluated by closed kinetic chain upper extremity stability test (CKCUEST). Shoulder internal and external rotation flexibility of the participants was evaluated with the shoulder joint internal and external rotation flexibility of motion test.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed athlete in a professional water polo team and actively participating in competitions
* Be between the ages of 10-25.
* Both genders

Exclusion Criteria:

* Having suffered an injury in the last 6 months
* Have any orthopedic, neurological, cardiovascular or any other health condition that prevents working in the last 6 months.
* Have a body mass index of 30 and above.
* Having undergone orthopedic surgery

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Flexibility | two weeks
  Shoulder Joint Internal and External Flexibility of Motion Test was used, from a standing position, the participant was asked to reach the lowest possible point of the back, over the shoulder, towards the floor, with the fingers extended and the palm facing the back, with external rotation of the arm. Then, he/she was asked to reach the highest point on his/her back by internal rotation, with the palm facing forward and again with the fingers in extension. The thoracic 5th vertebral process was used as the reference point to assess internal rotation motion and the cervical 7th vertebral process was used as the reference point to assess external rotation motion. If the thumb was not touching the reference point, the distance in cm was recorded as (-), if it was touching the reference point (0) and if it crossed the reference point, the distance in cm was recorded as (+).
Stability | two weeks
  Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), is a clinical test that measures the neuromuscular control of the upper extremity for shoulder stability. For the test, two bands were placed on the floor approximately 91.4 cm (36 inches) apart and parallel to the body of the subject. The test was performed in the push-up position. First, the subjects were asked for a few trial repetitions. Then, within 15 seconds, they were asked to quickly switch one hand to the other and each switch was recorded. After the test was repeated three times, the average of the recorded values was taken as the basis.
Strength | two weeks
  Shoulder strength was measured with a Cybex Humac Norm (Cybex, Lumex Inc. Division, Ronkonkoma, NY, USA) isokinetic dynamometer at angular velocities of 60°/s and 180°/s with a concentric/concentric protocol in the 90° abduction and external rotation position with the elbow fixed at 90° flexion. After a warm-up of 5 repetitions after the isokinetic dynamometer measured the end of gravitational correction and range of motion, the participant was asked to perform maximum internal rotation and external rotation, respectively, against the machine at 60°/s angular velocity for a total of 10 repetitions. The same procedure was then repeated for 15 repetitions at 180°/s angular velocity. This procedure was performed on both shoulders, dominant and non-dominant.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No